CLINICAL TRIAL: NCT04927585
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Polyvalent Env (A,B,C,A/E) / Gag (C) DNA and gp120 (A,B,C,A/E) Protein HIV-1 Vaccines (PDPHV-201401) Co-administered With or Without Adjuvant GLA-SE in Repeated Doses, in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of Polyvalent DNA/gp120 HIV Vaccine in Healthy, HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Worcester HIV Vaccine (Industry)
Collaborators: Brigham and Women's Hospital (Other); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WHV138
Record Dates: First submitted 2021-05-29; First posted 2021-06-16 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Genes, env; Vaccines, DNA; Plasmids; HIV Envelope Protein gp120; glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Treatment): DNA Vaccine + Protein Vaccine/GLA-SE (Experimental): Participants will receive 2 mg of env (A,B,C,A/E)/gag (C) DNA vaccine and 400 mcg of gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant at Day 0, and Months 3, 6, and 12.
  Interventions: Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine; Biological: gp120 (A,B,C,A/E) Protein Vaccine; Biological: GLA-SE adjuvant
- Group 1 (Control) (Placebo Comparator): Participants will receive placebo at Day 0, Months 3, 6, and 12.
  Interventions:
  Interventions: Biological: Placebo
- Group 2 (Treatment): Admixture of DNA Vaccine and Protein Vaccine (Experimental): Participants will receive admixture of 2 mg of env (A,B,C,A/E)/gag (C) DNA vaccine and 400 mcg of gp120 (A,B,C,A/E) protein vaccine (no adjuvant) at Day 0, and Months 1, 3, 6, and 8.
  Interventions: Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine; Biological: gp120 (A,B,C,A/E) Protein Vaccine
- Group 2 (Control) (Placebo Comparator): Participants will receive placebo at Day 0, and Months 1, 3, 6, and 8.
  Interventions:
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine — Administered by intramuscular injection in the deltoid
  Other Names: Polyvalent DNA (PDPHV-201401) Plasmid
  Arms: Group 1 (Treatment): DNA Vaccine + Protein Vaccine/GLA-SE; Group 2 (Treatment): Admixture of DNA Vaccine and Protein Vaccine
Biological: gp120 (A,B,C,A/E) Protein Vaccine — Administered by intramuscular injection in the deltoid
  Other Names: PDPHV-201401 Recombinant Proteins gp120A, gp120B, gp120C, gp120AE
  Arms: Group 1 (Treatment): DNA Vaccine + Protein Vaccine/GLA-SE; Group 2 (Treatment): Admixture of DNA Vaccine and Protein Vaccine
Biological: GLA-SE adjuvant — Administered by intramuscular injection in the deltoid.
  Other Names: glucopyranosyl lipid adjuvant-stable emulsion
  Arms: Group 1 (Treatment): DNA Vaccine + Protein Vaccine/GLA-SE
Biological: Placebo — Sodium Chloride for Injection, USP 0.9%; Administered by intramuscular injection in the deltoid.
  Arms: Group 1 (Control); Group 2 (Control)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and immunogenicity of polyvalent env (A,B,C,A/E)/gag (C) DNA and gp120 (A,B,C,A/E) protein vaccines (PDPHV201401) co-administered together with or without adjuvant in repeated doses in healthy, HIV-uninfected adults

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety, tolerability, and immunogenicity of polyvalent env (A,B,C,A/E)/gag (C) DNA and gp120 (A,B,C,A/E) protein vaccines (PDPHV201401) co-administered together with or without adjuvant in repeated doses in healthy, HIV-uninfected adults.

Participants will be enrolled in either Group 1 or 2 with Group 1 being enrolled first to compensate for the longer duration of vaccination period. Within each group, participants will be randomly assigned to either Treatment or Control.

Participants in Group 1 (Treatment) will receive polyvalent env (A,B,C,A/E)/gag (C) DNA vaccine in one arm and polyvalent gp120 (A,B,C,A/E) protein vaccine mixed with GLA-SE adjuvant in the other arm on Day 0 and at Months 3, 6, and 12. Participants in Group 1 (Control) will receive placebo on Day 0 and at Months 3, 6, and 12.

Participants in Group 2 (Treatment) will receive a mixture of polyvalent env (A,B,C,A/E)/gag (C) DNA vaccine and polyvalent gp120 (A,B,C,A/E) protein vaccine (without GLA-SE adjuvant) divided into two doses and administered into each arm on Day 0 and at Months 1, 3, 6, and 8. Participants in Group 2 (Control) will receive placebo on Day 0 and at Months 1, 3, 6, and 8.

Study visits for participants in Group 1 will occur on Day 0, Week 2, Months 3, 3.5, 6, 6.5, 12, 12 + 1 Week, 12.5, 18, and 24. Study visits for participants in Group 2 will occur on Day 0, Week 2, Months 1, 1.5, 3, 3.5, 6, 6.5, 8, 8 + 1 Week, 8.5, 14, and 20. Visits may include physical examination, blood and urine collection, HIV testing, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 50 years
2. Access to BWH trial site and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Agrees not to enroll in another study of an investigational research agent
6. Good general health as shown by medical history, physical exam, and screening laboratory tests
7. Willingness to receive HIV test results
8. Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
9. Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit. HVTN low risk guidelines will be used.

   Laboratory Inclusion Values Hemogram/CBC
10. Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 12.0 g/dL for volunteers who were born male
11. White blood cell count = 3,000 to 12,000 cells/mm3
12. Total lymphocyte count > 800 cells/mm3
13. Remaining differential either within institutional normal range or with site physician approval
14. Platelets = 125,000 to 450,000/mm3 Chemistry
15. Chemistry panel: ALT, AST, and alkaline phosphatase < 1.25 times the institutional upper limit of normal; creatinine < 1.1 times the institutional upper limit of normal.

    Virology
16. Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA).
17. Negative Hepatitis B surface antigen (HBsAg)
18. Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

    * Negative urine glucose, and
    * Negative or trace urine protein, and
    * Negative, trace, or 1+ urine hemoglobin (if 1+ hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

    Reproductive Status
19. Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
20. Reproductive status: A volunteer who was born female must:

    * Agree to consistently use effective contraception (see Appendix A and Appendix B) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until after the last required protocol clinic visit. Effective contraception is defined as using the following methods:

      * Condoms (male or female) with or without a spermicide,
      * Diaphragm or cervical cap with spermicide,
      * Intrauterine device (IUD),
      * Hormonal contraception, or
      * Any other contraceptive method approved by the PSRT
      * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy);
    * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
    * Or be sexually abstinent.
21. Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

1. Blood products received within 120 days before first vaccination
2. Investigational research agents received within 30 days before first vaccination
3. Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
4. Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing
5. Pregnant or breastfeeding
6. Active duty and reserve US military personnel Vaccines and other Injections
7. HIV vaccine(s) received in a prior HIV vaccine trial.
8. Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial, unless the vaccine subsequently received regulatory approval or emergency authorization.
9. Live attenuated vaccines, other than influenza vaccine, received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
10. Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
11. Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination Immune System
12. Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical immunosuppressives; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.)
13. Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
14. Immunoglobulin received within 60 days before first vaccination
15. Autoimmune disease, connective tissue disease, or history of vasculitis, eg, leukocytoclastic vasculitis, Henoch-Schonlein Purpura
16. Immunodeficiency Clinically significant medical conditions
17. Untreated or incompletely treated syphilis infection
18. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated injections or blood draws,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
    * Any condition specifically listed among the exclusion criteria below.
19. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
20. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
21. Current anti-tuberculosis (TB) prophylaxis or therapy
22. Asthma exclusion criteria:

    Asthma other than mild, well-controlled asthma.

    Exclude a volunteer who:
    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
    * In the past year has either of the following:
    * Greater than 1 exacerbation of symptoms treated with oral/ parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma
23. Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
24. Thyroidectomy, or thyroid disease requiring medication during the last 12 months
25. Hypertension:

    * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
    * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
26. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
27. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
28. Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
29. Asplenia: any condition resulting in the absence of a functional spleen
30. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Frequency of local injection site (including DTH) reactogenicity signs and symptoms | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Frequency of systemic reactogenicity signs and symptoms | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Frequency of adverse events (AEs) | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  AEs categorized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class, MedDRA preferred term, severity, and assessed relationship to study products
Severity of local injection site (including DTH) reactogenicity signs and symptoms | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Severity of systemic reactogenicity signs and symptoms | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Severity of adverse events (AEs) | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  AEs categorized by MedDRA system organ class, MedDRA preferred term, severity, and assessed relationship to study products
Number of participants with early discontinuation of vaccinations | Measured through participants' last study visit, at Month 20 to 24, depending on which part of the study participants are enrolled in
  Tabulated by reason and treatment arm

SECONDARY OUTCOMES:
Magnitude of serum HIV-1 Env-specific IgG responses | Measured at 2 weeks after the last vaccination
  Assessed by ELISA or Binding Antibody Multiplex Assay
Serum neutralizing antibody responses against Tier 1A, Tier 1B, and selected Tier 2 viruses | Measured at 2 weeks after the last vaccination
  Assessed by TZM-bl assay
Breadth of gp70-V1V2 IgG and gp120 IgA | Measured at 2 weeks after the last vaccination
  Assessed by ELISA or Binding Antibody Multiplex Assay, and ADCC activities against HIV-1 subtypes A, B, C and A/E
Frequency of HIV-1 specific CD4+ and CD8+ T-cell responses | Measured at 2 weeks after the last vaccination
  Assessed by intracellular cytokine staining (ICS)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No